CLINICAL TRIAL: NCT07407517
Title: Standard Chemotherapy Plus Oral Everolimus as Adjuvant Therapy for LAR Breast Cancer Patients: A Randomized, Open-Label, Phase III Trial （POLARIS）
Brief Title: Adjuvant Intensification for LAR
Acronym: POLARIS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of the Department of Breast Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N0108
Record Dates: First submitted 2026-01-14; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Females; Triple Negative Breast Cancer (TNBC)
Keywords: breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC-everolimus (Experimental): After completion of standard chemotherapy, everolimus at a fixed dose of 10 mg orally once daily continuously for a duration of 1 year.
  Interventions: Drug: Everolimus 10 mg daily
- SOC (No Intervention): After completion of standard chemotherapy, undergo observation and follow-up.

INTERVENTIONS:
Drug: Everolimus 10 mg daily — After completion of standard chemotherapy, everolimus at a fixed dose of 10 mg orally once daily continuously for a duration of 1 year.
  Arms: SOC-everolimus

SUMMARY:
This study enrolled patients with early-stage triple-negative breast cancer who had undergone radical surgery. The postoperative pathology met the TNM staging criteria of pT1c-3N0-3M0, and immunohistochemistry (IHC) results confirmed ER-negative status (IHC showed <1% of tumor cells positive for ER), PR-negative status (IHC showed <1% of tumor cells positive for PR), and HER2-negative status (IHC intensity of 0 or 1+; or IHC intensity of 2+ but with negative in situ hybridization results). Additionally, patients either exhibited high AR expression (IHC showing AR ≥10%) or were classified as the LAR subtype based on digital pathology.

This study plans to prospectively enroll 904 subjects, who will be randomized in a 1:1 ratio after completing standard chemotherapy. They will be allocated to either the standard-of-care (SOC) chemotherapy followed by everolimus group or the SOC-alone group. The study aims to evaluate the efficacy of SOC chemotherapy followed by everolimus versus SOC chemotherapy alone as adjuvant therapy for patients with early-stage radically resected triple-negative breast cancer of the LAR subtype, with the primary endpoint being 3-year invasive disease-free survival (iDFS).

ELIGIBILITY:
Inclusion Criteria:

-

Patients must meet **all** of the following inclusion criteria to be enrolled in this study:

1. Female, aged ≥18 years and ≤70 years.
2. ECOG performance status 0-1.
3. Histologically confirmed invasive triple-negative breast cancer (**definition**: breast cancer with estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER2) all confirmed negative by pathology. Specifically: **ER-negative**: IHC <1%; **PR-negative**: IHC <1%; **HER2-negative**: IHC 0/1+ or IHC 2+ but FISH/CISH negative. Additionally, histology must confirm **high AR expression**: AR IHC ≥10%, **or** digital pathology indicates the LAR subtype.
4. Underwent radical surgery for early-stage breast cancer, with postoperative pathology meeting TNM staging **pT1c-3N0-3M0**.
5. Patients with early-stage breast cancer who have received **at least 4 cycles of neoadjuvant chemotherapy containing anthracycline or taxane agents**, **did not achieve pathological complete response (pCR)**, and **do not carry pathogenic/likely pathogenic germline BRCA1/2 mutations**.
6. Adequate organ function, meeting the following criteria:

   * **Hematology**: HB ≥ 90 g/L (no transfusion within 14 days); ANC ≥ 1.5 × 10⁹/L; PLT ≥ 75 × 10⁹/L.

     * **Biochemistry**: TBIL ≤ 1.5 × ULN; ALT and AST ≤ 3 × ULN; serum Cr ≤ 1 × ULN, with creatinine clearance >50 mL/min (Cockcroft-Gault formula).
7. Surgical wound fully healed before study initiation.
8. Females of childbearing potential must use a medically approved contraceptive method during the study treatment and for at least 3 months after the last dose of study drug.
9. The patient voluntarily agrees to participate, signs the informed consent form, demonstrates good compliance, and agrees to follow-up.

Exclusion Criteria:

* Patients who meet **any** of the following criteria will be excluded from this study:

  1. Bilateral breast cancer.
  2. Metastatic disease at any site.
  3. Patients with cT > 2 cm or positive lymph nodes **and** carrying pathogenic/likely pathogenic germline BRCA1/2 mutations.
  4. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction within the past 6 months, or ventricular arrhythmia.
  5. History of clinically significant pulmonary disease, including but not limited to interstitial pneumonia, pneumonia, pulmonary fibrosis, and radiation pneumonitis (except for asymptomatic radiation changes not requiring intervention); or suspected such disease based on screening examinations.
  6. History of other malignancies within the past 5 years, excluding cured carcinoma in situ of the cervix, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
  7. Pregnant or lactating women; women of childbearing potential who cannot practice effective contraception.
  8. Patients concurrently participating in other clinical trials.
  9. Patients with a history of hypersensitivity or known allergy to any component of the study drugs; or patients with a history of allergy to other monoclonal antibodies.
  10. Severe or uncontrolled infection.
  11. Hypertension that cannot be adequately controlled with antihypertensive medication (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg).
  12. History of gastrointestinal bleeding within the past 6 months, or clear tendency for gastrointestinal bleeding, such as esophageal varices at risk of bleeding, locally active ulcerative lesions, or fecal occult blood ≥ (++). Patients with fecal occult blood (+) must undergo gastroscopy for further evaluation.
  13. Known active HBV or HCV infection (HBV-DNA ≥ 500 IU/mL), or chronic infection with abnormal liver function.
  14. Urinalysis showing urine protein ≥ ++, or 24-hour urine protein quantification > 1.0 g.
  15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to study enrollment.
  16. History of drug abuse (psychoactive substances) with inability to abstain, or history of psychiatric disorders.
  17. Patients deemed unsuitable for participation by the investigator's judgment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2033-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
iDFS | 3 year
  It is defined as the percentage of patients who remain free of invasive disease recurrence, secondary primary invasive cancers, or death from any cause over a 3-year period from randomization or initiation of study treatment.

SECONDARY OUTCOMES:
DFS | 3 year
  It measures the proportion of patients who remain free of detectable disease (including recurrence, progression, or new primary cancer) and alive for 3 years after starting treatment or randomization.
DDFS | 3year
  3-year DDFS is an oncology clinical trial endpoint that specifically measures the proportion of patients who remain free of distant metastasis (spread of cancer to remote organs) and death from the cancer within 3 years after initiation of study treatment or randomization. It focuses exclusively on distant metastatic events rather than all disease recurrences.
RFS | 3 year
  3-year RFS is an oncology clinical trial endpoint that measures the proportion of patients who remain free of disease recurrence (local, regional, or distant) for 3 years following curative-intent treatment (typically surgery). It specifically focuses on recurrence of the original primary cancer and does not include new primary cancers unrelated to the initial diagnosis.
OS | 3 year
  Overall Survival (OS) is the gold standard efficacy endpoint in oncology clinical trials, defined as the time from randomization (or treatment initiation) to death from any cause. It represents the most objective and clinically meaningful measure of treatment benefit, directly reflecting whether a therapy prolongs patients' lives.
Safety and Tolerability | 3 year
  Safety and Tolerability Will be Assessed According to Standard (CTCAE Version 5.0) Toxicity Reporting Criteria.
Quality of Life score in the per-protocol population | 3 year
  The quality of life of patients was assessed using the EORTC QLQ-C30 questionnaire before, during, and after treatment.

IPD SHARING:
Plan to Share IPD: No